CLINICAL TRIAL: NCT00808288
Title: A Phase 2b, Parallel Group, Placebo And Active Comparator Controlled Study To Investigate The Safety, Toleration And Efficacy Of 6-Week Once Daily Administration Of Inhaled PF-00610355 Dry Powder In Patients With Moderate Chronic Obstructive Pulmonary Disease.
Brief Title: A Study To Investigate The Safety, Toleration And Efficacy of PF00610355 In Chronic Obstructive Pulmonary Disease (COPD) Patients.
Acronym: A7881013
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A7881013
Record Dates: First submitted 2008-12-12; First posted 2008-12-15 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Lung Diseases; Lung Diseases, Obstructive
Keywords: COPD Respiratory Long acting beta agonist
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases; Lung Diseases, Obstructive | interventions — N-((4'-hydroxybiphenyl-3-yl)methyl)-2-(3-(2-((-2-hydroxy-2-(4-hydroxy-3-((methylsulfonyl)amino)phenyl)ethyl)amino)-2-methylpropyl)phenyl)acetamide; Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- PF-00610355 (Experimental)
  Interventions: Drug: PF-00610355
- PF- 00610355 (Experimental)
  Interventions: Drug: PF - 00610355
- PF - 00610355 (Experimental)
  Interventions: Drug: PF- 00610355
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Salmeterol (Active Comparator)
  Interventions: Drug: Salmeterol

INTERVENTIONS:
Drug: PF-00610355 — oral, inhaled, dry powder, 600ug, OD
  Arms: PF-00610355
Drug: PF - 00610355 — oral, inhaled, dry powder, 300ug, OD
  Arms: PF- 00610355
Drug: PF- 00610355 — oral, inhaled, dry powder, 100ug, OD
  Arms: PF - 00610355
Drug: Placebo — oral, inhaled, dry powder, placebo, OD
  Arms: Placebo
Drug: Salmeterol — salmeterol, 50ug, BID
  Arms: Salmeterol

SUMMARY:
To assess the effects and safety of PF-00610355 on patients with chronic obstructive lung disease (COPD)

ELIGIBILITY:
Inclusion Criteria:

* Post-bronchodilator FEV1/FVC ratio <0.7 and a post-bronchodilator FEV1 of 50-80%.
* Diagnosis of moderate COPD for a minimum of 6 months.
* Stable disease for at least 1 month prior to screening

Exclusion Criteria:

* More than 2 exacerbations of COPD requiring treatment with oral steroids in the preceding year or hospitalisation for the treatment of COPD within 3 months of screening or more than twice during the preceding year.
* History of a lower respiratory tract infection or significant disease instability during the month preceding screening or during the time between screening and randomisation.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2010-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in trough FEV1 | 6 week

SECONDARY OUTCOMES:
Maximal and mean changes from baseline in heart rate, QTc and plasma potassium | each visit
Change from baseline in peak FEV1 | 0-6 hours /6 weeks
Change from baseline in trough and peak FEV6, FVC and IC | 6 weeks
Change from baseline in trough FEV1, FEV6, forced vital capacity (FVC) and inspiratory capacity (IC) | 2 and 4 weeks
Change from baseline in Respiratory Questionnaire Self-Administered Standardised (CRQ-SAS) | 2,4,6 weeks
Change from baseline of COPD symptoms and rescue bronchodilator use (per daily diary). | weekly

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (67):
- United States (25):
  - Pfizer Investigational Site, Fairhope, Alabama
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Spring Valley, California
  - Pfizer Investigational Site, Wheat Ridge, Colorado
  - Pfizer Investigational Site, Daytona Beach, Florida
  - Pfizer Investigational Site, Ormond Beach, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Trinity, Florida
  - Pfizer Investigational Site, Austell, Georgia
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Fridley, Minnesota
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, Rochester, Minnesota
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Lincoln, Rhode Island
  - Pfizer Investigational Site, Pawtucket, Rhode Island
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Columbia, South Carolina
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Morgantown, West Virginia
- Argentina (2):
  - Pfizer Investigational Site, Rosario, Santa Fe Province
  - Pfizer Investigational Site, Buenos Aires
- Bulgaria (4):
  - Pfizer Investigational Site, Rousse
  - Pfizer Investigational Site, Sofia
  - Pfizer Investigational Site, Stara Zagora
  - Pfizer Investigational Site, Troyan Municipality
- Pfizer Investigational Site, Zagreb, Croatia
- Czechia (4):
  - Pfizer Investigational Site, Kutná Hora
  - Pfizer Investigational Site, Liberec
  - Pfizer Investigational Site, Prague
  - Pfizer Investigational Site, Tábor
- Germany (7):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Frankfurt
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, Kassel
  - Pfizer Investigational Site, Lübeck
  - Pfizer Investigational Site, Schwerin
  - Pfizer Investigational Site, Wiesbaden
- Hungary (5):
  - Pfizer Investigational Site, Budapest
  - Pfizer Investigational Site, Debrecen
  - Pfizer Investigational Site, Szeged
  - Pfizer Investigational Site, Szombathely
  - Pfizer Investigational Site, Törökbálint
- Poland (4):
  - Pfizer Investigational Site, Lodz
  - Pfizer Investigational Site, Sopot
  - Pfizer Investigational Site, Warsaw
  - Pfizer Investigational Site, Wejherowo
- Slovakia (6):
  - Pfizer Investigational Site, Bojnice
  - Pfizer Investigational Site, Bratislava
  - Pfizer Investigational Site, Liptovský Hrádok
  - Pfizer Investigational Site, Nové Zámky
  - Pfizer Investigational Site, Poprad
  - Pfizer Investigational Site, Spišská Nová Ves
- South Africa (5):
  - Pfizer Investigational Site, Bellville, Cape Town
  - Pfizer Investigational Site, Tygerberg, Cape Town
  - Pfizer Investigational Site, Bloemfontein, Free State
  - Pfizer Investigational Site, Bloemfontein
  - Pfizer Investigational Site, Gatesville, Cape Town
- Spain (2):
  - Pfizer Investigational Site, Salt, Girona
  - Pfizer Investigational Site, Pozuelo de Alarcón, Madrid
- Turkey (Türkiye) (2):
  - Pfizer Investigational Site, Istanbul
  - Pfizer Investigational Site, Izmir

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7881013&StudyName=A%20Study%20To%20Investigate%20The%20Safety%2C%20Toleration%20And%20Efficacy%20of%20PF00610355%20In%20Chronic%20Obstructive%20Pulmonary%20Disease%20%28COPD%29%20Patients.